CLINICAL TRIAL: NCT06033547
Title: A Phase I, Open-label, Single Dose Escalation Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Two Different Formulations of Long-acting Cabotegravir Administered to Healthy Adult Participants
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Two Different Formulations of Long-acting Cabotegravir in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 219406
Expanded Access: NCT03462810 (Available)
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections
Keywords: Cabotegravir; Pharmacokinetics
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Participants receiving Cabotegravir Formulation F (Experimental)
  Interventions: Drug: Cabotegravir Formulation F
- Part B: Participants receiving Cabotegravir Formulation G (Experimental)
  Interventions: Drug: Cabotegravir Formulation G

INTERVENTIONS:
Drug: Cabotegravir Formulation F — Cabotegravir Formulation F will be administered
  Arms: Part A: Participants receiving Cabotegravir Formulation F
Drug: Cabotegravir Formulation G — Cabotegravir Formulation G will be administered
  Arms: Part B: Participants receiving Cabotegravir Formulation G

SUMMARY:
The primary purpose of the study is to investigate the safety, tolerability, and pharmacokinetic (PK) profiles of two different cabotegravir formulations in healthy adult participants. The study will initially start with the assessment of Cabotegravir Formulation F. Once the clinical batch of Cabotegravir Formulation G is available, this formulation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight =>40 kilogram (kg) and body mass index (BMI) within the range =>18 to =<32 kilogram per meter square (kg/m^2)
* Participants who are negative on a single test for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)(approved molecular polymerase chain reaction [PCR] laboratory or point of care test) performed on the day of admission. A negative result is required prior to the administration of study intervention on Day 1.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Participants assigned female at birth are eligible to participate if they are not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a woman of childbearing potential (WOCBP) OR
* Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1% from the time of screening and inclusive of the entire time while on the study.
* A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within the 30 days before the first dose of study intervention.
* Capable of giving written informed consent

Exclusion Criteria:

* Current presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities.
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including participants who have required treatment for seizures within this time period.
* Participants who in the investigator's judgment, poses a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* Positive SARS-CoV-2 polymerase chain reaction test, having signs and symptoms which in the opinion of the investigator are suggestive of COVID-19 (i.e., fever, cough etc) within 14 days of inpatient admission, or having contact with known COVID-19 positive person/s in the 14 days prior to inpatient admission.
* Human immunodeficiency virus (HIV-1 or HIV-2) infection as indicated by positive antibody/antigen test.
* History of or on-going high-risk behaviors that, in the opinion of the investigator, may put the participant at increased risk for HIV infection including, but not limited to, participants in HIV discordant relationships, or men who report current or prior unprotected anal sex with other men and those reporting prior or current injecting drug use.
* Presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* Abnormal blood pressure.
* Evidence of previous myocardial infarction.
* Any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular [AV] block [2nd degree or higher], Wolff- Parkinson-White [WPW] syndrome).
* Any significant arrhythmia which, in the opinion of the investigator or the medical monitor, will interfere with the safety for the individual participant.
* One or more exclusionary values for a screening Electrocardiogram (ECG).
* Alanine transaminase (ALT) >1.5x upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Estimated Glomerular Filtration Rate (eGFR) <60 milliliter per minute (mL/min) using the Chronic Kidney Disease - Improved Prediction Equations (CKD-EPI) Creatinine Equation (2021).
* Haemoglobin <12.5 gram per deciliter (g/dL) for men and <11 g/dL for women.
* Positive pre-study drug/alcohol screen.
* Regular use of tobacco- or nicotine-containing products within 3 months prior to screening; or urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g., nicotine patches or vaporizing devices).
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for males or >7 units for females.
* Regular use of known drugs of abuse.
* Concurrent participation in another clinical trial (except imaging trials); or has participated in a clinical trial and received an investigational product within the following time period prior to the first dosing day in this study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than four (4) new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study interventions (or components thereof), a history of drug allergy or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation
* Current or anticipated need for chronic anti-coagulation therapy (with the exception of low-dose aspirin =< 325 mg/day)
* Hereditary coagulation and platelet disorders (e.g., haemophilia or Von Willebrand disease [VWD]).
* Participant has a tattoo overlying the location of injection or an underlying skin disease or condition (e.g., infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) that, in the opinion of the investigator, may interfere with interpretation of injection site reactions or administration of study intervention.
* Any other clinical condition, behaviour or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study; unable to comply with dosing requirements; or unable to comply with study visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of cabotegravir | Up to Week 52
Time of maximum observed plasma concentration (tmax) of cabotegravir | Up to Week 52
Area under the concentration - time curve from time zero to 4 weeks following the injection (AUC[0-4]) of cabotegravir | Up to Week 4
Plasma Concentration of cabotegravir at Week 4 | Week 4
Number of participants with adverse events (AEs) based on severity | Up to Week 52
Absolute value of haematology parameter: Platelet count (cells per microliter) | Up to Week 52
Absolute value of haematology parameter: Red Blood Cell Count (RBC) (million cells per microliter) | Up to Week 52
Absolute values of haematology parameters: haemoglobin (Hgb) (grams per decilitre) | Up to Week 52
Absolute values of haematology parameters: haematocrit (Proportion of red blood cells in blood) | Up to Week 52
Absolute value of haematology parameter: Mean Corpuscle Volume (MCV) (Femtoliters) | Up to Week 52
Absolute value of haematology parameter: Mean Corpuscle haemoglobin (MCH) (Picograms) | Up to Week 52
Absolute values of haematology parameters: Reticulocytes (Percentage of reticulocytes) | Up to Week 52
Absolute values of haematology parameters: Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per litre) | Up to Week 52
Absolute values of Clinical Chemistry parameters: Glucose (fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per decilitre) | Up to Week 52
Absolute values of Clinical Chemistry parameters: AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per litre) | Up to Week 52
  Clinical chemistry parameters such as Aspartate Aminotransferase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase and (SGPT), Alkaline phosphatase (ALP) and Creatinine Phosphokinase (CPK) will be analysed.
Absolute values of Clinical chemistry parameters: Total Protein (Grams per deciliter) | Up to Week 52
Absolute values of Clinical chemistry parameters: Estimated Glomerular Filtration Rate (eGFR2) (millilitres per minute) | Up to Week 52
Change from Baseline in haematology parameter: Platelet count (cells per microliter) | Baseline (Day 1) and up to Week 52
Change from Baseline in haematology parameter: Red Blood Cell Count (RBC) (million cells per microliter) | Baseline (Day 1) and up to Week 52
Change from baseline in haematology parameters: haematocrit (Proportion of red blood cells in blood) | Baseline (Day 1) and up to Week 52
Change from baseline in haematology parameter: Mean Corpuscle Volume (MCV) (Femtoliters) | Baseline (Day 1) and up to Week 52
Change from baseline in haematology parameter: Mean Corpuscle haemoglobin (MCH) (Picograms) | Baseline (Day 1) and up to Week 52
Change from baseline in haematology parameters: Reticulocytes (Percentage of reticulocytes) | Baseline (Day 1) and up to Week 52
Change from baseline in haematology parameters: Differential count of Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils (giga cells per litre) | Baseline (Day 1) and up to Week 52
Change from baseline in Clinical Chemistry parameters: Glucose (fasting), Blood Urea Nitrogen (BUN), Creatinine, Sodium, Potassium, Calcium, Direct Bilirubin and Total Bilirubin (milligrams per decilitre) | Baseline (Day 1) and up to Week 52
Change from baseline in Clinical Chemistry parameters: AST/SGOT, ALT/ SGPT, ALP and CPK (International Units per litre) | Baseline (Day 1) and up to Week 52
  Clinical chemistry parameters such as Aspartate Aminotransferase (AST) / Serum Glutamic-Oxaloacetic Transaminase (SGOT), Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase and (SGPT), Alkaline phosphatase (ALP) and Creatinine Phosphokinase (CPK) will be analysed
Change from baseline in Clinical chemistry parameters: Total Protein (Grams per deciliter) | Baseline (Day 1) and up to Week 52
Change from baseline in Clinical chemistry parameters: Estimated Glomerular Filtration Rate (eGFR) (millilitres per minute) | Baseline (Day 1) and up to Week 52

SECONDARY OUTCOMES:
Area under the concentration - time curve from time zero to infinity (AUC[0-inf]) of cabotegravir | Up to Week 52
Area under the concentration - time curve from time zero to time of last quantifiable concentration [AUC(0-last)] of cabotegravir | Up to Week 52
Plasma Concentration of cabotegravir at Week 8,12 and 24 | Week 8, 12 and 24
Apparent terminal phase half-life (t1/2) of cabotegravir | Up to Week 52
Apparent long-acting absorption rate constant (KA-LA) of cabotegravir | Up to Week 52
Dose proportionality of cabotegravir based on AUC(0-inf), AUC(0-last), Cmax, and plasma concentration (Unit of measure: Slope of log dose) | Up to Week 52
Number of participants with maximum post-baseline QTc values compared to baseline by category (to <=450 milliseconds (msec) or no change, to >450 msec to <=480 msec, to >480 msec to <=500 msec, and to >500 msec) | Up to Week 52
Number of participants with maximum post-baseline increase in QTc values compared to baseline based on category (increase <=30 msec, increase of 31-60 msec, and increase of >60 msec) | Up to Week 52
Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline for diastolic blood pressure (DBP), systolic blood pressure (SBP) and pulse rate | Up to Week 52
  Number of participants with worst case post-baseline values relative to potential clinical importance criteria compared to baseline will be categorized into change to low, change to within range or no change, and change to high

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/